CLINICAL TRIAL: NCT04681729
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Parallel-group Study of Dupilumab in Patients With Chronic Inducible Cold Urticaria Who Remain Symptomatic Despite the Use of H1-antihistamine Treatment
Brief Title: Dupilumab for the Treatment of Chronic Inducible Cold Urticaria in Patients Who Remain Symptomatic Despite the Use of H1-antihistamine (LIBERTY-CINDU CUrIADS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16720; 2020-003756-33 (EudraCT Number); U1111-1246-6913 (Registry Identifier: ICTRP)
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09-02

CONDITIONS: Cold Urticaria
MeSH Terms: conditions — Cold Urticaria | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab (Experimental): Dose regimens, on top of regular or as needed non-sedating H1-antihistamine
  Interventions: Drug: Dupilumab SAR231893; Drug: Non sedating H1-antihistamine
- Matched Placebo (Placebo Comparator): Placebo, on top of regular/as needed non-sedating H1-antihistamine
  Interventions: Drug: Placebo; Drug: Non sedating H1-antihistamine

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form: Injection solution Route of administration: Subcutaneous
  Arms: Dupilumab
Drug: Placebo — Pharmaceutical form: Injection solution Route of administration: Subcutaneous
  Arms: Matched Placebo
Drug: Non sedating H1-antihistamine — Pharmaceutical form: Tablet Route of administration: Oral

SUMMARY:
Primary Objective:

To demonstrate the efficacy of dupilumab in adult and adolescent participants with primary acquired chronic inducible cold urticaria (ColdU) who remain symptomatic despite the use of an H1-antihistamine

Secondary Objectives:

To demonstrate the efficacy of dupilumab on primary acquired chronic inducible ColdU disease control To demonstrate the efficacy of dupilumab on primary acquired chronic inducible ColdU local signs and symptoms (hives/wheals, itch, burning sensation and pain) after provocation test To demonstrate the efficacy of dupilumab on primary acquired chronic inducible ColdU disease activity To demonstrate improvement in health-related quality-of-life and overall disease status and severity To evaluate the ability of dupilumab in reducing the proportion of participants who require rescue therapy To evaluate the proportion of participants with cold exposure triggered urticaria To evaluate safety outcome measures To evaluate immunogenicity of dupilumab

DETAILED DESCRIPTION:
The duration of study for each participant included 2-4 weeks of screening period, 24 weeks of treatment period and 12 weeks of post treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participant had to be ≥12 years to 80 years of age inclusive at the time of signing the informed consent
* Participants who had a diagnosis of primary acquired chronic inducible ColdU defined as recurrence of itchy wheals and/or angioedema due to cold for longer than 6 weeks prior to screening visit (Visit 1)
* Participants with positive ice cube provocation test, ie, presenting at least a confluent hive/wheal on the exposed skin area, at the screening visit (Visit 1) and randomization visit (Visit 2)
* Participants meeting at least 1 of the following criteria despite regular/daily or as needed use of H1-antihistamine (AH):

  * Urticaria Control Test (UCT) (4 item) <12 at the screening visit (Visit 1) and randomization visit (Visit 2)
  * Within 6 months prior to the screening visit, documented medical history of cold exposure triggered anaphylaxis or oropharyngeal edema
  * Within 6 months prior to the screening visit, documented medical history of cold exposure triggered urticaria requiring emergency medical care visit or treatment with epinephrine
* Participants using a study defined H1-antihistamine regularly/daily or as needed for primary acquired chronic inducible cold urticaria
* Body weight ≥30 kg

Exclusion Criteria:

Participants were excluded from the study if any of the following criteria applied:

* Clearly defined underlying etiology for urticaria other than primary acquired chronic inducible ColdU
* Presence of skin morbidities other than cold urticaria that may interfere with the assessment of the study outcomes
* Active atopic dermatitis
* Severe concomitant illness(es) that, in the investigator's judgment, would have adversely affected the patient's participation in the study
* Active tuberculosis or non-tuberculous mycobacterial infection, or a history of incompletely treated tuberculosis unless documented adequately treated.
* Diagnosed active endoparasitic infections; suspected or high risk of endoparasitic infection
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals within 2 weeks before the screening visit and during the screening period
* Known or suspected immunodeficiency
* Active malignancy or history of malignancy within 5 years before the baseline visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin
* History of systemic hypersensitivity or anaphylaxis to any other biologic therapy or any of its excipients.
* Participation in prior dupilumab clinical study, or have been treated with commercially available dupilumab.

The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (33):
- United States (5):
  - Allergy and Asthma Medical Group and Research Center-Site Number:8400001, San Diego, California
  - Treasure Valley Medical Research-Site Number:8400007, Boise, Idaho
  - Allergy & Asthma Specialists, PSC-Site Number:8400003, Owensboro, Kentucky
  - Johns Hopkins University (Asthma and Allergy Center)-Site Number:8400005, Baltimore, Maryland
  - Bernstein Allergy Group Inc-Site Number:8400004, Cincinnati, Ohio
- Argentina (6):
  - Investigational Site Number :0320001, CABA, Buenos Aires
  - Investigational Site Number :0320005, CABA, Buenos Aires
  - Investigational Site Number :0320006, CABA, Buenos Aires
  - Investigational Site Number :0320002, Rosario, Santa Fe Province
  - Investigational Site Number :0320004, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number :0320003, Buenos Aires
- Canada (9):
  - Investigational Site Number :1240008, Edmonton, Alberta
  - Investigational Site Number :1240010, Edmonton, Alberta
  - Investigational Site Number :1240007, Hamilton, Ontario
  - Investigational Site Number :1240009, Hamilton, Ontario
  - Investigational Site Number :1240001, Toronto, Ontario
  - Investigational Site Number :1240011, Montreal, Quebec
  - Investigational Site Number :1240005, Saint-Charles-Borromée, Quebec
  - Investigational Site Number :1240006, Sherbrooke, Quebec
  - Investigational Site Number :1240002, Québec
- Germany (6):
  - Investigational Site Number :2760002, Berlin
  - Investigational Site Number :2760004, Dresden
  - Investigational Site Number :2760007, Erlangen
  - Investigational Site Number :2760006, Hanover
  - Investigational Site Number :2760005, Leipzig
  - Investigational Site Number :2760001, Mainz
- Japan (7):
  - Investigational Site Number :3920002, Nagoya, Aichi-ken
  - Investigational Site Number :3920003, Hiroshima, Hiroshima
  - Investigational Site Number :3920008, Kamimashiki Gun, Kumamoto
  - Investigational Site Number :3920007, Sakai-shi, Osaka
  - Investigational Site Number :3920010, Koto-ku, Tokyo
  - Investigational Site Number :3920011, Tachikawa-shi, Tokyo
  - Investigational Site Number :3920009, Habikino-Shi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16720 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25251&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 32 active sites in 5 countries. A total of 123 participants were screened between 10 December 2020 and 22 June 2022, of which 41 were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 82 participants were randomized in 1:1 ratio to receive the study treatment with dupilumab or placebo. Randomization was stratified by age (adults versus adolescents with body weight [BW] greater than or equal to [>=] 60 kilograms [kg] or >=30 kg and less than [<] 60 kg), country and background H1-antihistamine regular/daily use (Yes/No).
Groups:
- Placebo: Participants based on their BW >=60 kg or BW >=30 kg and <60 kg received loading dose of placebo (matched to dupilumab 600 milligrams [mg] or 400 mg) subcutaneous (SC) injection on Day 1, respectively, followed by placebo (matched to dupilumab 300 mg or 200 mg) SC injection every 2 weeks (q2w) up to Week 22 along with their established standard of care background therapy with a long-acting non-sedating H1- antihistamine.
- Dupilumab: Participants based on their BW >=60 kg or >=30 kg and <60 kg received loading dose of dupilumab 600 mg or 400 mg SC injection on Day 1, respectively, followed by dupilumab 300 mg or 200 mg SC injection q2w up to Week 22 along with their established standard of care background therapy with a long-acting non-sedating H1-antihistamine.
Period: Overall Study
Arm/Group | Placebo | Dupilumab
Started | 40 | 42
Completed | 30 | 31
Not Completed | 10 | 11
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 8 | 9

BASELINE CHARACTERISTICS:
Population: Randomized population consisted of all participants from the screened population who had been allocated to randomized intervention by interactive response technology regardless of whether the treatment kit was used or not.
Groups:
- Placebo: Participants based on their BW >=60 kg or BW >=30 kg and <60 kg received loading dose of placebo (matched to dupilumab 600 mg or 400 mg) SC injection on Day 1, respectively, followed by placebo (matched to dupilumab 300 mg or 200 mg) SC injection q2w up to Week 22 along with their established standard of care background therapy with a long-acting non-sedating H1- antihistamine.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (16.3) | 33.0 (13.1) | 35.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 63
  Male | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 35 | 35 | 70
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Negative Ice Cube Provocation Test at Week 24
Description: The ice cube provocation test is the most frequently used provocation method for cold urticaria (ColdU). A negative ice cube provocation test was defined as the absence of confluent hives/wheal at the entire skin site of exposure after ice cube provocation test. Ice cube was applied on forearm skin for 5 minutes. Provocation test reading time was 10 minutes after removal of ice cube.
Time Frame: Week 24
Population: The Intent-to-treat (ITT) population consisted of all randomized participants who had been allocated to a randomized intervention by IRT regardless of whether the treatment kit was used or not and were analyzed according to the intervention group allocated by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
percentage of participants | 37.5 | 40.5
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; A hierarchical testing procedure was used to control the family-wise type-I error. Testing was then performed sequentially in order the endpoints were reported and continued when primary endpoint was statistically significant at two-sided 0.01; Test type: Superiority; p = 0.9492, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test was performed on the association between the ice cube provocation test result and intervention group, stratified by region and background H1-antihistamine regular/daily use (Yes or No). Threshold of significance at 0.01; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.41 to 2.56]

2. Secondary Outcome: Change From Baseline in Urticaria Control Test (UCT) Scale Scores at Week 24
Description: UCT is validated patient reported outcome (PRO) questionnaire used for assessing urticaria control. UCT has been developed and validated with participants Chronic Spontaneous Urticaria (CSU) and Chronic inducible urticaria (CIndU). It comprised of 4 items: severity of physical symptoms of urticaria (itch, hives and/or swelling); quality of life (QoL) impairment; frequency of treatment being not sufficient to control urticaria; overall urticarial control. Each item was rated on a 5-point Likert scale ranged from 0 (high disease activity) to 4 (low disease activity). The UCT total score was calculated as sum of all 4 individual item scores,ranged from 0 to 16. Higher scores indicated low disease activity, complete disease control, and vice-versa. Least square (LS) mean and standard error (SE) were analyzed using Analysis of covariance (ANCOVA) model with corresponding Baseline value, intervention group, region and background H1-antihistamine regular/daily use (Yes or No) as covariates.
Time Frame: Baseline to Week 24
Population: The ITT population consisted of all randomized participants who had been allocated to a randomized intervention by IRT regardless of whether the treatment kit was used or not and were analyzed according to the intervention group allocated by randomization. Only data from the participants analyzed were reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 30 | 32
score on a scale | 3.75 (0.89) | 4.36 (0.80)

3. Secondary Outcome: Percentage of Participants With Urticaria Control Test Score >=12 at Week 24
Description: The UCT is a validated PRO questionnaire used for assessing urticaria control. The questionnaire has been developed and validated with participants with CSU and CIndU. It comprised of 4 items: severity of physical symptoms of urticaria (itch, hives and/or swelling); QoL impairment; frequency of treatment being not sufficient to control urticaria; overall urticarial control. Each item was rated on a 5-point Likert scale ranging from 0 to 4, with low score indicating high disease activity and low disease control, and vice-versa. The UCT total score was calculated as sum of all 4 individual item scores, which ranged from 0 to 16. Higher scores indicated low disease activity and complete disease control, and vice-versa. A score of >=12 on the scale indicates well-controlled urticaria. Percentage of participants with UCT score >=12 (i.e., well controlled urticaria) at Week 24 are reported in this endpoint.
Time Frame: Week 24
Population: The ITT population consisted of all randomized participants who had been allocated to a randomized intervention by IRT regardless of whether the treatment kit was used or not and were analyzed according to the intervention group allocated by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
percentage of participants | 27.5 | 33.3

4. Secondary Outcome: Percentage of Participants With an Improvement of >=3 Points From Baseline in Urticaria Control Test Score at Week 24
Description: The UCT is a validated PRO questionnaire used for assessing urticaria control. The questionnaire has been developed and validated with participants with CSU and CIndU. It comprised of 4 items: severity of physical symptoms of urticaria (itch, hives and/or swelling); QoL impairment; frequency of treatment being not sufficient to control urticaria; overall urticarial control. Each item was rated on a 5-point Likert scale ranging from 0 (high disease activity) to 4 (low disease activity), with low score indicating high disease activity and low disease control, and vice-versa. The UCT total score was calculated as sum of all 4 individual item scores, which ranged from 0 to 16. Higher scores indicated low disease activity and complete disease control, and vice-versa.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
percentage of participants | 30.0 | 45.2

5. Secondary Outcome: Change From Baseline in Local Wheal Intensity Likert Scale Score at Weeks 12 and 24
Description: Wheal intensity Likert scale (ranging from 0 to 5) is a clinician-reported endpoint completed at the study visit, 10 minutes after removal of the ice cube from the participants' arm. The scale comprised of a single item assessing the intensity of participants' cutaneous reaction rated as follows: 0 = no wheals; 1 = numerous small, non-coalescent wheals; 2 = a large, regular, slightly edematous, coalescent wheal; 3 = a large and moderately edematous wheal; 4 = a large, regular, and significantly edematous wheal without pseudopodia; and 5 = a large, very edematous wheal with pseudopodia. Higher score indicated greater severity. LS mean and SE were analyzed using ANCOVA model with the corresponding Baseline value, intervention group, region and background H1-antihistamine regular/daily use (Yes or No) as covariates.
Time Frame: Baseline, Week 12 and Week 24
Population: The ITT population consisted of all randomized participants who had been allocated to a randomized intervention by IRT regardless of whether the treatment kit was used or not and were analyzed according to the intervention group allocated by randomization. Here, only participants with available data for each specified category were reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
score on a scale
  Week 12: number analyzed (Participants) | 38 | 39
  Week 12 | -1.49 (0.23) | -1.19 (0.23)
  Week 24: number analyzed (Participants) | 32 | 33
  Week 24 | -1.52 (0.28) | -1.55 (0.27)

6. Secondary Outcome: Change From Baseline in Local Itch Severity Scale Score at Weeks 12 and 24
Description: Local itch (pruritus) severity was assessed using the peak pruritus numerical rating scale (NRS). Peak pruritus NRS is a PRO comprised of a single item rated on a scale ranged from 0 ("No itch") to 10 ("Worst itch imaginable"), where higher scores indicated worse itch. Participants were asked to rate the intensity of their worst local site itch (pruritus) 10 minutes after removal of the ice cube. LS mean and SE were analyzed using ANCOVA model with the corresponding Baseline value, intervention group, region and background H1-antihistamine regular/daily use (Yes or No) as covariates.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
score on a scale
  Week 12: number analyzed (Participants) | 35 | 34
  Week 12 | -2.12 (0.58) | -2.52 (0.59)
  Week 24: number analyzed (Participants) | 30 | 29
  Week 24 | -2.18 (0.63) | -2.43 (0.62)

7. Secondary Outcome: Change From Baseline in Local Skin Burning Sensation Scale Score at Weeks 12 and 24
Description: Local skin burning sensation was assessed using peak burning sensation NRS which is a PRO comprised of a single item rated on a scale ranged from 0 ("No burning sensation") to 10 ("Worst imaginable burning sensation"). Higher score indicated worst burning sensation. Participants were asked to rate the intensity of the worst local site burning sensation of their skin 10 minutes after the removal of the ice cube. LS mean and SE were analyzed using ANCOVA model with the corresponding Baseline value, intervention group, region and background H1-antihistamine regular/daily use (Yes or No) as covariates.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
score on a scale
  Week 12: number analyzed (Participants) | 35 | 34
  Week 12 | -1.60 (0.60) | -2.43 (0.61)
  Week 24: number analyzed (Participants) | 30 | 29
  Week 24 | -1.76 (0.69) | -2.04 (0.68)

8. Secondary Outcome: Change From Baseline in Local Pain Severity Scale Score at Weeks 12 and 24
Description: Local pain severity was assessed using peak pain NRS. The peak pain NRS is a PRO comprised of a single item rated on a scale ranged from 0 ("No pain") to 10 ("Worst imaginable pain"). Higher score indicated worst pain. Participants were asked to rate the intensity of their worst local site pain 10 minutes after removal of the ice cube. LS mean and SE was analyzed using ANCOVA model with the corresponding Baseline value, intervention group, region and background H1-antihistamine regular/daily use (Yes or No) as covariates.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
score on a scale
  Week 12: number analyzed (Participants) | 35 | 34
  Week 12 | -1.82 (0.54) | -2.14 (0.55)
  Week 24: number analyzed (Participants) | 30 | 29
  Week 24 | -1.60 (0.58) | -2.28 (0.57)

9. Secondary Outcome: Percentage of Participants With Negative Ice Cube Provocation Test at Week 12
Description: The ice cube provocation test is the most frequently used provocation method for ColdU. A negative ice cube provocation test was defined as the absence of confluent hives/wheal at the entire skin site of exposure after ice cube provocation test. Ice cube was applied on forearm skin for 5 minutes. Provocation test reading time was 10 minutes after removal of ice cube.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
percentage of participants | 35.0 | 31.0

10. Secondary Outcome: Change From Baseline in Cold Urticaria Signs and Symptoms Severity Scale Score at Week 24
Description: Cold Urticaria Activity Score (ColdUAS) is disease-specific PRO questionnaire designed to determine cold urticaria disease activity. Intended for participants with cold urticaria aged 12 years old and above; developed and comprehensively tested with adults and adolescent participants with cold urticaria. Disease activity assessment was based on daily documentation of cold-induced skin reactions (wheals and swelling), skin sensations (itching, burning, pain or feeling hot), avoidance behavior and trigger exposure, and overall symptoms severity. Skin reaction, skin sensations, exposition to cold temperatures that usually cause ColdU symptoms and overall symptom severity were rated on a 4-point scale ranged from 0 (less severe) to 4 (more severe), where higher score indicated more signs and symptoms. LS mean and SE were analyzed using ANCOVA model with corresponding Baseline value, intervention group, region and background H1-antihistamine regular/daily use (Yes/No) as covariates.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 24
score on a scale | -1.04 (0.23) | -1.28 (0.22)

11. Secondary Outcome: Change From Baseline in Percentage of Cold Urticaria Sign and Symptom-Free Days at Week 24
Description: ColdUAS: disease-specific PRO questionnaire to determine cold urticaria disease activity in adults and adolescents with cold urticaria. For change from Baseline in percentage of cold urticaria sign and symptom-free days, responses to ColdUAS question (Q) 1 (rating severity of signs: wheals and swelling) and ColdUAS, Q2 (rating severity of symptoms: itch, burning, pain, or feeling hot) on days exposed to cold (ColdUAS Q3 responded Yes) were used. Within 14-day interval before each visit the number of sign and symptom-free days (ColdUAS Q1=0 and Q2=0) on days exposed to cold (ColdUAS Q3 greater than >0) was counted and divided by total number of days exposed to cold in this interval. Percentage of cold urticaria sign and symptom free days = sign and symptom free days/cold exposure days in 14 days window*100. LS mean and SE by ANCOVA model with the corresponding Baseline value, intervention group, region and background H1-antihistamines regular/daily use (Yes/No) as covariates.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 24
percentage of days | 15.66 (7.49) | 27.82 (7.26)

12. Secondary Outcome: Change From Baseline in Health-related Quality-of-life (HRQoL) as Measured by Dermatology Life Quality Index (DLQI) Scale Scores at Week 24
Description: DLQI is a PRO developed to measure dermatology-specific HRQoL in adults. It comprises 10 items assessing the impact of skin disease on participant's HRQoL over the previous week. The items cover symptoms, leisure activities, work/school or holiday time, personal relationships including intimate, side effects of treatment, and emotional reactions to having a skin disease. It is a validated questionnaire used in clinical practice and clinical trials. For 9-items; response scale was a 4-point Likert scale ranging from 0 = "Not at all" to 3 = "Very much", where higher score=more impact of QoL, and vice-versa. The remaining 1 item about work/studying was rated on a 3-point Likert scale ranged from 0="Not at all" to 2="A lot". DLQI total score was the sum of score of all the items and ranged from 0 to 30, with a high score indicated poor HRQoL, and vice-versa. LS mean and SE from ANCOVA model.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 28 | 29
score on a scale | -4.70 (1.08) | -4.32 (1.00)

13. Secondary Outcome: Change From Baseline in Cold Urticaria Quality of Life (ColdU-QoL) Scale Score at Week 24
Description: The ColdU-QoL questionnaire is a disease-specific PRO questionnaire designed to assess the impact of cold urticaria on participant's HRQoL. It has been developed and comprehensively tested with adults and adolescent participants with cold urticaria. The questionnaire contains 19 items, each rated using a 5-point Likert scale ranged from 0 (Not at all / Never) to 4 (Very much / Very often). The total raw score of the ColdU-QoL was transformed to a 0 to 100 score for analysis using the formula: ColdU-QoL total score = Sum of the score of all completed items/Maximum possible sum of the score of all completed items*100. Higher scores indicated higher ColdU-related QoL impairment, and vice-versa. LS mean and SE were analyzed from ANCOVA model with the corresponding Baseline value, intervention group, region and background H1-antihistamine regular/daily use (Yes or No) as covariates.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 31 | 32
score on a scale | -20.12 (3.81) | -20.07 (3.65)

14. Secondary Outcome: Percentage of Participants Receiving Rescue Therapy for Primary Acquired Chronic Inducible Cold Urticaria
Description: Rescue therapy included additional doses of H1-antihistamines and short course of oral corticosteroids (OCS).
Time Frame: From first investigational medicinal product (IMP) administration (Day 1) up to Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
percentage of participants
  H1-antihistamines | 32.5 | 45.2
  OCS | 2.5 | 0

15. Secondary Outcome: Percentage of Participants With Cold Exposure Triggered Urticaria That Required Hospitalization/Emergency Medical Care Visit or Treatment With Epinephrine
Description: Percentage of participants with cold exposure triggered urticaria that required hospitalization/emergency medical care visit or treatment with epinephrine are reported in this endpoint.
Time Frame: From first IMP administration (Day 1) up to 14 weeks after last IMP administration (i.e., up to Week 36)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 40 | 42
percentage of participants
  Hospitalization/emergency medical care visit | 0 | 0
  Epinephrine treatment | 0 | 0

16. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Serious adverse events (SAEs) was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the treatment-emergent period (from the first IMP administration to the last IMP administration + 14 weeks).
Time Frame: From first IMP administration (Day 1) up to 14 weeks after last IMP administration (i.e., up to Week 36)
Population: The Safety population consisted of all participants who were randomized and received at least 1 dose of IMP and were analyzed according to the intervention actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 39 | 43
Participants
  TEAEs | 27 | 23
  TESAEs | 0 | 1

17. Secondary Outcome: Number of Participants With Treatment-emergent Antidrug Antibodies (ADA) Response
Description: ADA response was categorized as: Treatment-emergent and Treatment-boosted. Treatment-emergent ADAs were defined as a positive response in the ADA assay post-first dose, when baseline results were negative or missing. Treatment-boosted ADAs: defined as an ADA positive response in the assay post first dose that was >=4-fold over baseline titer levels, when Baseline results were positive. Titer values were defined as low titer (< 1,000); moderate (1,000 less than or equal to [<=] titer <=10,000) and high titer (> 10,000).
Time Frame: From first IMP administration (Day 1) up to 14 weeks after last IMP administration (i.e., up to Week 36)
Population: The ADA population consisted of all participants who were randomized and received at least 1 dose of IMP and had at least 1 non-missing ADA result after first dose of IMP. Participants were analyzed according to the intervention actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 36 | 38
Participants
  Treatment-emergent ADAs | 0 | 4
  Treatment-boosted ADAs | 0 | 0

ADVERSE EVENTS:
Time Frame: From first IMP administration (Day 1) up to 14 weeks after last IMP administration (i.e., up to Week 36)
Description: The Safety population consisted of all participants who were randomized and received at least 1 dose of IMP and were analyzed according to the intervention actually received.
Groups:
- Placebo: Participants based on their BW >=60 kg or BW >=30 kg and <60 kg received loading dose of placebo (matched to dupilumab 600 mg or 400 mg) SC injection on Day 1, respectively, followed by placebo (matched to dupilumab 300 mg or 200 mg) SC injection q2w up to Week 22 along with their established standard of care background therapy with a long-acting non-sedating H1-antihistamine.
Arm/Group | Placebo | Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/43
Other Adverse Events (participants affected / at risk) | 16/39 | 14/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | Dupilumab (N=43)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | Dupilumab (N=43)
Injection Site Erythema (General disorders) | 0 (0) | 3 (4)
Injection Site Pain (General disorders) | 1 (1) | 4 (8)
Injection Site Reaction (General disorders) | 1 (1) | 6 (26)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Covid-19 (Infections and infestations) | 8 (8) | 5 (5)
Suspected Covid-19 (Infections and infestations) | 3 (3) | 2 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT04681729/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT04681729/SAP_001.pdf